CLINICAL TRIAL: NCT03583216
Title: Comparison of Factor XII Levels in Gestational Diabetic and Healthy Pregnancies
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Esra Ozbasli, Ass. Prof., Acibadem University
Other Study IDs: ATADEK-2017/10
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Diabetic Pregnancy; Pregnancy Related; Complement System; Disorder
Keywords: Diabetic pregnancies, Factor XII
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 8ml of blood samples will be drawn from each participitant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic pregnancy: Pregnant patients with a diagnosis of Type I, Type II or gestational diabetes will be included in this arm. Blood will be drawn from each patient when they are hospitalized and before they deliver either vaginally or by cesarean section. Blood will be drawn into two citrate tubes, each will contain 4 ml blood.
  Interventions: Diagnostic Test: Diabetic pregnancy
- Non-diabetic pregnancy: Healthy non-diabetic pregnant patients will be included in this arm. Blood will be drawn from each patient when they are hospitalized and before they deliver either vaginally or by cesarean section. Blood will be drawn into two citrate tubes, each will contain 4 ml blood.
  Interventions: Diagnostic Test: Non-diabetic pregnancy

INTERVENTIONS:
Diagnostic Test: Diabetic pregnancy — Blood samples will be drawn before delivery to evaluate Factor XII level.
  Groups: Diabetic pregnancy
Diagnostic Test: Non-diabetic pregnancy — Blood samples will be drawn before delivery to evaluate Factor XII level.
  Groups: Non-diabetic pregnancy

SUMMARY:
To compare Factor XII levels in gestational diabetic and healthy pregnancies.

DETAILED DESCRIPTION:
Thirty singleton term pregnant women with a diagnosis of Type I, Type II or gestational diabetes and thirty singleton uncomplicated term healthy pregnant women will be included in our study. Our study will be performed at Istanbul Acibadem Maslak Hospital, Turkey. Blood will be drawn from each patient when they are hospitalized and before they deliver either vaginally or by cesarean section. Blood will be drawn into two citrate tubes, each will contain 4 ml blood. Blood will be transferred to the lab immediately and will be centrifuged. The supernatant will be stored at -80°C. When the anticipated number of samples are completed Factor XII levels will be calculated in each sample.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy
* Pregnant patients with a diagnosis of Type I diabetes
* Pregnant patients with a diagnosis of Type II diabetes
* Pregnant patients with a diagnosis of Gestational diabetes
* Non-diabetic pregnancies
* Uncomplicated pregnancies

Exclusion Criteria:

* Preterm pregnancy
* Postterm pregnancy
* Pregnant patients with a diagnosis of systemic diseases other than diabetes
* Complicated pregnancies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: 30 Pregnant patients with a diagnosis of Type I, Type II or gestational diabetes and 30 non-diabetic pregnant patients will be included in our trial.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Factor XII level | Blood will be drawn when the patient is hospitalized before they deliver.
  The primary outcome is to evaluate Factor XII level in diabetic pregnancies. If the investigators can prove that Factor XII, which has a mitogenic activity and can increase the risk for thrombosis, increases more in diabetic pregnancies in the future usage of Factor inhibitors may reduce macrosomia, thrombosis and the complications due to these conditions in diabetic pregnancies

SECONDARY OUTCOMES:
Macrosmia | Blood will be drawn when the patient is hospitalized before they deliver.
  The secondary outcome is to prove that the increase of Factor XII level is higher diabetic pregnancies and this increase might have an effect on macrosomia.

CONTACTS AND LOCATIONS:
Overall Officials: Mete Gungor, Prof., Study Director — Acibadem MAA University
Locations (1):
- Acibadem Maslak Hospital, Istanbul, Sariyer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Background] Schousboe I. Pharmacological regulation of factor XII activation may be a new target to control pathological coagulation. Biochem Pharmacol. 2008 Mar 1;75(5):1007-13. doi: 10.1016/j.bcp.2007.10.003. Epub 2007 Oct 7. PMID 17996217
- [Background] Decrem Y, Rath G, Blasioli V, Cauchie P, Robert S, Beaufays J, Frere JM, Feron O, Dogne JM, Dessy C, Vanhamme L, Godfroid E. Ir-CPI, a coagulation contact phase inhibitor from the tick Ixodes ricinus, inhibits thrombus formation without impairing hemostasis. J Exp Med. 2009 Oct 26;206(11):2381-95. doi: 10.1084/jem.20091007. Epub 2009 Oct 5. PMID 19808248
- [Background] Bryant JW, Shariat-Madar Z. Human plasma kallikrein-kinin system: physiological and biochemical parameters. Cardiovasc Hematol Agents Med Chem. 2009 Jul;7(3):234-50. doi: 10.2174/187152509789105444. PMID 19689262
- [Result] Renne T, Schmaier AH, Nickel KF, Blomback M, Maas C. In vivo roles of factor XII. Blood. 2012 Nov 22;120(22):4296-303. doi: 10.1182/blood-2012-07-292094. Epub 2012 Sep 19. PMID 22993391
- [Derived] Ozbasli E, Takmaz O, Karabuk E, Gungor M. Comparison of factor XII levels in gestational diabetes, fetal macrosomia, and healthy pregnancies. BMC Pregnancy Childbirth. 2020 Dec 2;20(1):752. doi: 10.1186/s12884-020-03455-0. PMID 33267793